CLINICAL TRIAL: NCT03277989
Title: INFINITY™Total Ankle Replacement Follow-up
Acronym: ITAR
Status: Terminated | Type: Observational
Why Stopped: Business Decision
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: US17-TAR-001
Record Dates: First submitted 2017-09-08; First posted 2017-09-11 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
Study Title INFINITY™Total Ankle Replacement Follow-up (ITAR) Study Design Prospective, multi-site, multi-year post-market clinical follow-up study Study Group Primary/Unilateral and/or bilateral Total Ankle Arthroplasty subjects implanted with INFINITY™ Total Ankle System Number of Subjects 150 with 9 sites

DETAILED DESCRIPTION:
The primary outcome measure of this post-market clinical observational study is to collect data relating to the INFINITY™ Total Ankle System survivorship at 10 years. The secondary outcome measures are to characterize the improvements after implantation over a 10 year period using patient reported outcome measures related to quality of life, pain and functional improvements, safety of the implants, as well as radiographic assessments (X-Rays)

The outcome measures collected in this study will be analyzed and reported as required for local, regional, and country requirements (i.e., regulatory authorities and notified bodies).

ELIGIBILITY:
Inclusion Criteria:

* Be 21 years of age or older at the time of surgery;
* Diagnosed with unilateral and/or bilateral ankle joint disease;
* Diagnosed with ankle joint damage from rheumatoid arthritis, post-traumatic, or degenerative arthritis;
* Willing and able to consent to participate (written, informed consent;
* Willing and able to attend the requested follow-up visits;
* A clinical decision has been made to use INFINITY™ Total Ankle System replacement prior to enrollment in the research.

Exclusion Criteria:

* Subjects with an ankle condition, as determined by the investigator, to be an inappropriate candidate for a total ankle replacement;
* Subjects requiring revision total ankle replacement of the ankle being considered for study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary/Unilateral and/or bilateral Total Ankle Arthroplasty subjects implanted with INFINITY™ Total Ankle System
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gibson, Study Director — Stryker Trauma and Extremities
Locations (9):
- United States (9):
  - Eisenhower Medical Center, Rancho Mirage, California
  - Orthopaedic & Spine Center of the Rockies, Fort Collins, Colorado
  - Illinois Bone & Joint Institute, Libertyville, Illinois
  - Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan
  - Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Slocum Center for Orthopedics & Sports Medicine, Eugene, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Erlanger, Chattanooga, Tennessee
  - Campbell Clinic, Germantown, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- INFINITY™ Total Ankle System: Study subjects included those withankle joints damaged by severe rheumatoid arthritis, post-traumatic disease, and degenerative arthritis and implanted with the INFINITY™ Total Ankle System.
Period: Overall Study
Arm/Group | INFINITY™ Total Ankle System
Started | 155
Completed | 0
Not Completed | 155
Not completed — Lost to Follow-up | 6
Not completed — Adverse Event | 6
Not completed — Withdrawal by Subject | 3
Not completed — Didn't Receive Study Device | 7
Not completed — Site Closure | 26
Not completed — Sponsor Closure | 107

BASELINE CHARACTERISTICS:
Population: Of the 155 subjects enrolled, 148 received the study device and were therefore analyzed
Groups:
- INFINITY™ Total Ankle System: Study subjects included those with ankle joints damaged by severe rheumatoid arthritis, post-traumatic disease, and degenerative arthritis and implanted with the INFINITY™ Total Ankle System.
Arm/Group | INFINITY™ Total Ankle System
Number analyzed (Participants) | 148
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1
  Race: Hispanic | 1
  Race: Multi-racial | 0
  Race: White | 139
  Race: Other | 7
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.03 (5.17)
Smoking Status [Count of Participants; unit: Participants]
  Never | 94
  Previous | 50
  Current, <= 1 Pack/day | 4
Primary Diagnosis [Count of Participants; unit: Participants]
  Degenerative Arthritis | 72
  Rheumatoid Arthritis | 4
  Post Traumatic Arthritis | 71
  Other | 1

OUTCOME MEASURES:

1. Primary Outcome: Survivorship at 10 Years
Description: The primary endpoint is a survivorship rate at 10 years as defined with a Kaplan Meier survivorship analysis.
Time Frame: 10 years
Population: Since the study was prematurely discontinued where the maximum subject follow-up is two years, no survival analysis was conducted.
Arm/Group | INFINITY™ Total Ankle System
Number analyzed (Participants) | 0

2. Secondary Outcome: Radiographic Evaluation-physician Reported Questionnaire
Description: Identify and assess the implant for the below:
  Evidence of Subsidence Evidence Tibia and Talar Subsidence > 5° Evidence of Radiolucency Evidence Tibia and Talar Linear Radiolucency > 2mm and document if the Radiolucency is Progressive Evidence of Tibia and Talar Cystic Radiolucency > 5mm and document if the Radiolucency is Progressive Other Radiographic Findings deemed reportable by Investigator
Time Frame: Pre-op through 2 years
Measure: Count of Participants; unit: Participants
Groups:
- INFINITY™ Total Ankle System at 2 Years: Study subjects included those with ankle joints damaged by severe rheumatoid arthritis, post-traumatic disease, and degenerative arthritis and implanted with the INFINITY™ Total Ankle System.
Arm/Group | INFINITY™ Total Ankle System at 2 Years
Number analyzed (Participants) | 115
Participants
  No Radiographic Finding | 80
  Any Evidence of Radiolucency < 2mm linear and <5mm cystic radiolucency | 20
  Other | 10
  Subsidence | 2
  Tibia: linear radiolucency > 2mm | 2
  Talus: linear radiolucency > 2mm | 1
  Tibia: linear radiolucency Progressive | 0
  Talus: linear radiolucency Progressive | 0
  Talus: cystic radiolucency > 5mm | 0
  Tibia: cystic radiolucency > 5mm | 0
  Talus: cystic radiolucency Progessive | 0
  Tibia: cystic radiolucency Progessive | 0
  Tibia Subsidence >5 | 0
  Talus Subsidence >5 | 0

3. Secondary Outcome: PROMIS Scale v1.2- Global Health
Description: PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates andmonitors physical, mental, and social health in adults and children. It can be used with the general population and with individuals living with chronic conditions. (PROMIS Scale v1.2- Global Health) The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. The results of the questions are used to calculate two summary scores: a Global Physical Health Score and a Global Mental Health score. These scores are then standardized to the general population, using the "T-Score". The average "TScore" for the United States population is 50 points, with a standard deviation of 10 points. Higher scores indicate a healthier patient. Will report change from baseline score to 2 years.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Total T-score
Arm/Group | INFINITY™ Total Ankle System at 2 Years
Number analyzed (Participants) | 116
Total T-score
  Total Global Physical Health | 50.9 (8.51)
  Total Global Mental Score | 53.4 (9.23)

4. Secondary Outcome: Ankle Osteoarthritis Score (AOS)
Description: AOS is a reliable, validated, visual analog-based, disease-specific self-administered instrument designed specifically to measure disability and pain from ankle osteoarthritis. Both Pain and Disability components are used to calculate the total score. The score is from zero to one hundred with a lower score indicating more normal function. A minimal clinically important difference (MCID) for the Total AOS score reduction from baseline has been established: 12.35 points. Will report change from baseline score to 2 years.
Time Frame: Pre-op though 2 years
Measure: Mean (Standard Deviation); unit: Change in score from baseline
Arm/Group | INFINITY™ Total Ankle System at 2 Years
Number analyzed (Participants) | 113
Change in score from baseline | -39 (21.2)

5. Secondary Outcome: FAOS Questionnaire
Description: The FAOS is a self-report measure that evaluates symptoms and functional limitations in individuals with generalized foot and ankle disorders. The FAOS is composed of the following 5 subscales: pain (9 items), other symptoms (7 items), activities of daily living (7 items), sports and recreational activities (5 items), and foot and ankle-related quality of life (4 items). All subscales have a range from 0 (severe symptoms) to 100 (no symptoms). The total FAOS score is calculated by summing up the scores from each of the five subscales (pain, other symptoms, activities of daily living, sports and recreation, and quality of life) after individually calculating each subscale score by adding up the points from its respective questions and dividing by the maximum possible score for that subscale; the final result is then normalized to a scale from 0 (severe symptoms) to 100 (no symptoms) based on the total score across all subscales. We report change from baseline score to 2 years.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | INFINITY™ Total Ankle System at 2 Years
Number analyzed (Participants) | 116
Scores on a Scale
  Total FAOS Score | 75.5 (18.6)
  Total Symptoms Score | 75.0 (20.4)
  Total Pain Score | 82.4 (18.7)
  Total Activities of Daily Living Score | 87.2 (16.7)
  Total Sport/Recreation Score | 63.2 (29.9)
  Total QOL Score | 69.1 (24.4)

6. Secondary Outcome: TAR Satisfaction Questionnaire
Description: Compare satisfaction of total ankle replacement post operatively utilizing a four point scale
Time Frame: Pre-op through 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | INFINITY™ Total Ankle System at 2 Years
Number analyzed (Participants) | 110
Participants
  Excellent | 81
  Good | 22
  Fair | 3
  Poor | 4

ADVERSE EVENTS:
Time Frame: Surgery to 5 years, 1 month, 13 days
Description: Procedural and device related events will be described and collected on the AE form. It is the responsibility of the operating surgeon/s to be aware and note the adverse effects from the package insert/instructions for use by the manufacturer/sponsor.
Arm/Group | INFINITY™ Total Ankle System
All-Cause Mortality (participants affected / at risk) | 0/148
Serious Adverse Events (participants affected / at risk) | 9/148
Other Adverse Events (participants affected / at risk) | 33/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFINITY™ Total Ankle System (N=148)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Periprosthetic osteolysis (Injury, poisoning and procedural complications) | 1 (1)
Ankle impingement (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Device loosening (Product Issues) | 2 (2)
Ankle arthroplasty (Surgical and medical procedures) | 1 (1)
Ankle operation (Surgical and medical procedures) | 1 (2)
Knee arthroplasty (Surgical and medical procedures) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFINITY™ Total Ankle System (N=148)
Complication associated with device (General disorders) | 1 (1)
Implant site hypoaesthesia (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2)
Stress fracture (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (14)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (6)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysaesthesia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Nerve compression (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Device loosening (Product Issues) | 1 (1)
Implant subsidence (Product Issues) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 1 (1)
Ankle arthroplasty (Surgical and medical procedures) | 1 (1)
Arthrotomy (Surgical and medical procedures) | 1 (1)
Cast application (Surgical and medical procedures) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As the study was terminated early, outcomes and adverse events can only be reported up to the date of closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-08-10): https://cdn.clinicaltrials.gov/large-docs/89/NCT03277989/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/89/NCT03277989/SAP_001.pdf